CLINICAL TRIAL: NCT04352972
Title: Innovative Tele-monitored Home-Based Program for Post Total Knee Replacement Rehabilitation: A Noninferiority Randomized Controlled Trial
Brief Title: Hospital-based Usual cAre Versus Tele-monitoring Rehabilitation
Acronym: HUATR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: University of the Sunshine Coast (Unknown); Duke University (Other); Duke-NUS Graduate Medical School (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TA18may-0007
Record Dates: First submitted 2020-04-10; First posted 2020-04-20 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the intervention, it is not feasible to blind participants or the treating physiotherapists. To reduce bias, the outcome assessor will be blinded to treatment allocation. Participants will also be instructed not to reveal details about their group assignment to the outcome assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-based rehabilitation program (Active Comparator)
  Interventions: Other: Hospital-based rehabilitation program
- Tele-monitored home exercise program (Experimental)
  Interventions: Device: Tele-monitored home exercise program

INTERVENTIONS:
Device: Tele-monitored home exercise program — Tele-monitoring home exercise program used in the home with monitoring by physiotherapists.
  Arms: Tele-monitored home exercise program
Other: Hospital-based rehabilitation program — Participants will receive a maximum of 8 sessions over 10 weeks with the option of two additional sessions. Participants will receive exercises, patient education, manual therapy and other modalities that were prescribed and progressed at the project physiotherapist's discretion. Participants will also receive a set of home exercises and they will be instructed to exercise on days when not attending rehabilitation.
  Arms: Hospital-based rehabilitation program

SUMMARY:
Knee osteoarthritis (OA) is a common, chronic, and costly condition, and patients with advanced knee OA and severe disability often require a total knee replacement (TKR) surgery. In Singapore, after TKR surgery, nearly all patients who are home discharged are referred to hospital-based outpatient rehabilitation. Although outpatient rehabilitation attendance is associated with better functional outcomes, access to rehabilitation care is limited as outpatient rehabilitation is costly and inconvenient for patients and their caregivers, resulting in suboptimal adherence. A tele-monitored home-based exercise program provides the best access to rehabilitation care and is a potential alternative for the majority of patients who do not require intensive "hands-on" rehabilitation therapy.

The primary aim of this non-inferiority randomized controlled trial is to compare patient functional outcomes and cost-effectiveness of an innovative tele-monitored rehabilitation program versus that of currently standard, hospital-based outpatient rehabilitation program among patients post TKR.

DETAILED DESCRIPTION:
Study Hypotheses

Primary hypothesis: A 10-week home-based exercise program, combined with tele-monitoring of functional outcomes, will not be inferior to an 10-week hospital-based rehabilitation at 3 and at 6 months after total knee replacement (TKR) in improving physical function (fast gait speed).

Secondary hypothesis 1: A 10-week home-based exercise program, combined with tele-monitoring of functional outcomes, will not be inferior to a 10-week hospital-based rehabilitation at 3 and at 6 months after TKR in improving knee pain, physical impairments, and health-related quality of life.

Secondary hypothesis 2: A 10-week tele-monitored home-based exercise program will be more cost-effective than the 10-week hospital-based rehabilitation in total TKR-related costs

Approach and Methods

This will be an assessor-blinded, parallel design, non-inferiority randomised controlled trial, with assessments preoperatively(baseline), 3 months, and 6 months after total knee replacement surgery. The protocol conforms to the CONSORT guidelines for non-inferiority randomized controlled trials. Post TKR, all participants will undergo daily inpatient rehabilitation. At discharge, they will be given a standard booklet with advice on ice therapy and home exercises to be performed. Two weeks post TKR, randomization will occur and participants will be randomised to receive either the telemonitored home exercise program or the hospital-based rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral total knee replacement
* Age >= 45 years
* Willingness to be randomized to either tele-monitored home exercise program or outpatient rehabilitation program
* Ability to provide informed consent

Exclusion Criteria:

* Further lower limb joint replacement surgery anticipated within the next 6 months
* Rheumatoid arthritis and other systemic arthritis
* A previous history of stroke and other major neurological conditions
* An intention to transfer to step-down care facilities post-operatively.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Difference in Fast-paced gait speed | Pre-operation; 3 months and 6 months post-surgery
  Difference in fast gait speed (over 10 metres) between the two treatment groups.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Pre-operation; 3 months and 6 months post-surgery
  The physical function subscale of the Knee injury and Osteoarthritis Outcome Score (KOOS) is designed to evaluate the patient's opinion about their physical function. All items are scored on 5-point Likert scales. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for the subscale.
Quadriceps muscle strength | Pre-operation; 3 months and 6 months post-surgery
  Maximum voluntary isometric torque of the quadriceps muscles (at 70 degrees knee flexion) will be measured using a Biodex dynamometer
30s chair stand test | Pre-operation; 3 months and 6 months post-surgery
  Total number of sit-to-stand repetitions completed in 30 seconds will be recorded. This is a measure of lower limb strength and endurance.
Knee Pain: Numeric Pain Rating Scale (NPRS) | Pre-operation; 3 months and 6 months post-surgery
  Knee pain intensity during climbing stairs, walking, and sitting-to-standing will be measured using separate 11-point numeric pain rating scale, with zero representing no pain at all and 10 representing worst imaginable pain.
Knee range-of-motion | Pre-operation; 3 months and 6 months post-surgery
  A long-arm goniometer will be used to measure active-assisted knee flexion and extension range-of-motion with the participants in supine position.
EuroQol-5 Dimensions (EQ-5D-5L) descriptive system | Pre-operation; 3 months and 6 months post-surgery
  The EuroQol-5 Dimensions (EQ-5D-5L) is a standardised instrument to measure health related quality of life in cost-effectiveness analysis. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patients' decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Cost | 3 months and 6 months post-surgery
  Cost questionnaire measuring the direct and indirect costs.
Treatment satisfaction: scale | 3 months post-surgery
  Participants will rate their satisfaction with treatment on a 11 point likert scale, with 0 indicating "no satisfaction" and 10 indicating "complete satisfaction".
Treatment credibility | 3 months post-surgery
  To assess participants' confidence about the benefits of the intervention. Participants will rate their satisfaction with treatment on a 11 point likert scale, with 0 indicating "not confident" and 10 indicating "extremely confident".
STarT Back Screening Tool | Pre-operation; 3 months and 6 months post-surgery
  The psychological subscale of the STarT Back Screening Tool will be determined by summing all items related to fear, anxiety, catastrophizing, depression, and bothersomeness. The STarT Back Screening Tool will be modified for use in the total knee replacement population by replacing the word "back" with "knee".
Örebro Musculoskeletal Pain Screening Questionnaire (short form) | Pre-operation; 3 months and 6 months post-surgery
  This 10 item questionnaire evaluates psychological factors that potentially influence pain and/or function. These items are scored 0-10, where 0 refers to absence of impairment and 10 to severe impairment. Three items need to be reversed in order for all the questions to be oriented in the same direction. The total score will range between 1 and 100. A score above 50 indicates higher estimated risk for future work disability.

OTHER OUTCOMES:
Number of adverse events | 3 months and 6 months post-surgery
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pua YH, Koh SS, Terluin B, Woon EL, Chew ES, Yeo SJ, Chen JY, Liow LMH, Clark R, Thumboo J. Effect of Context Specificity on Response to the Shortened WOMAC Function Scale in Patients Undergoing Total Knee Arthroplasty. Arch Phys Med Rehabil. 2024 Sep;105(9):1725-1732. doi: 10.1016/j.apmr.2024.05.005. Epub 2024 May 7. PMID 38723858